CLINICAL TRIAL: NCT02121951
Title: Quadratus Lumborum Block Versus Local Anesthetic Infiltration Combined With Monitored Anesthesia Care for Percutaneous Nephrostomy
Brief Title: Quadratus Lumborum Block for Percutaneous Nephrostomy
Acronym: QLB
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ghada M N Bashandy, Dr, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Quadratus Lumborum Block
Record Dates: First submitted 2014-04-20; First posted 2014-04-24 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Nephrostomy; Complications; Upper Urinary Tract Dilatation and Obstruction; Regional Anesthesia Morbidity; Adverse Anesthesia Outcome
Keywords: Percutaneous Nephrostomy; Quadtatus Lumborum Block; Cancer; Monitored Anaesthesia Care
MeSH Terms: conditions — Bites and Stings; Neoplasms | interventions — Lidocaine; Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Local Anesthetic infiltration and MAC (Active Comparator): * Local Anesthetic infiltration with 1% lignocaine
  * MAC with IV Midazolam Img\ml and Fentanyl 10 mic\ml
  Interventions: Procedure: Local Anesthetic infiltration; Drug: MAC
- Quadratus Lumborum block and MAC (Experimental): * QL block with 0.25% levobupivacaine (Chirocaine, Abbott, Ireland) and 1% lignocaine
  * MAC with IV Midazolam Img\ml and Fentanyl 10 mic\ml
  Interventions: Procedure: Quadratus Lumborum block; Drug: MAC

INTERVENTIONS:
Procedure: Local Anesthetic infiltration — Lignocaine infiltration through the nephrostomy track
  Other Names: Lignocaine
  Arms: Local Anesthetic infiltration and MAC
Procedure: Quadratus Lumborum block — A linear 12-MHz ultrasound probe will be placed in the anterior axillary line to visualize the typical triple abdominal layers. Then, the probe will be placed in the midaxillary line and at this point the layers of abdominal layers starte to taper. The probe will be placed in the posterior axillary line, sonoanatomy will show first the transversus abdominis disappearing then the internal oblique and external oblique forming aponeurosis and appearance of QL will be noticed. At the posterior border of the quadratus lumborum muscle and outside the fascia, Touhe needle will be inserted in plane and confirmed its position by injecting saline. Under ultrasound (US) guidance, local anesthetic mixure will be deposited separating the fascia
  Other Names: -0.25% levobupivacaine (Chirocaine, Abbott, Ireland); -1% lignocaine
  Arms: Quadratus Lumborum block and MAC
Drug: MAC — Incremental doses are given to the targed sedation and analgesia
  Other Names: -Midazolam: 1 mg\ml; -Fentanyl: 10 mic\ml

SUMMARY:
Percutaneous nephrostomy (PCN) is one of the interventions in the radiology department in which pain control is necessary. Quadratus Lumborum (QL) block will be tried to limit the use of systemic analgesics and its accompanying untoward effects in those frail patients requiring PCN that is performed in the prone position.

DETAILED DESCRIPTION:
Quadratus Lumborum block is a novel technique in which extension into the thoracic paravertebral space may occur. QL block would seem to be able to alleviate both somatic and visceral pain so it's expected to decrease the need for systemic sedation\analgesia to a minimum.

ELIGIBILITY:
Inclusion Criteria:

1. ASA grade III and IV patients,
2. Ureteral obstruction due to malignancy or secondary to urinary diversion after cystectomy

Exclusion Criteria:

1. Bleeding diathesis; INR more than than 1.5 and platelet count less than 100,000/mm3.
2. Untreated urinary tract infection;
3. Pre-operative haemoglobin <10 gm/dl,
4. Severely co morbid patients
5. Non-dilated renal collecting system
6. Patient refusal to consent for the procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Analgesia | 4 hours
  Verbal Rating Scale is assessed for degree of pain during the procedure and after till discharge from the radiology department.

SECONDARY OUTCOMES:
Respiratory Depression | 4 hours
  Respiratory rate and airway patency is monitored with an anesthesiologist.
Sedation | 4 hours
  Ramsay Seadation Score is assessed during and after procedure till discharge
Cardiovascular stability | 4 hours
  Blood pressure and Heart rate is assessed during and after procedure till discharge
Patient Satisfaction | 48 hours
  Patient Satisfaction Quistionaire

CONTACTS AND LOCATIONS:
Overall Officials: Dina N Abbas, M D, Study Director — National Cancer Institute, Egypt; Ghada M Bashandy, MD, Principal Investigator — National Cancer Institute, Egypt; Wael Darwish, M D, Study Chair — National Cancer Institute, Egypt
Locations (1):
- National Cancer Institute, Cairo, Old Cairo, Egypt

REFERENCES:
- [Result] Kadam VR. Ultrasound-guided quadratus lumborum block as a postoperative analgesic technique for laparotomy. J Anaesthesiol Clin Pharmacol. 2013 Oct;29(4):550-2. doi: 10.4103/0970-9185.119148. PMID 24249997
- [Result] Ironfield CM, Barrington MJ, Kluger R, Sites B. Are patients satisfied after peripheral nerve blockade? Results from an International Registry of Regional Anesthesia. Reg Anesth Pain Med. 2014 Jan-Feb;39(1):48-55. doi: 10.1097/AAP.0000000000000038. PMID 24310051